CLINICAL TRIAL: NCT02262884
Title: A Physician Preference Study of the Use of SurgiQuest AirSeal vs. Conventional Insufflation Systems for the Management of Pneumoperitoneum in Robotic Partial Nephrectomy .
Brief Title: SurgiQuest AirSeal in Robotic Partial Nephrectomy - (TARPAN Study)
Acronym: TARPAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SurgiQuest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRT DD112313
Record Dates: First submitted 2014-09-30; First posted 2014-10-13 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Subcutaneous Emphysema
MeSH Terms: conditions — Subcutaneous Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AIS @ 12mmHg pressure (Active Comparator): SurgiQuest AirSeal Insufflation System (AIS) set at 12mmHg pressure for the management of pneumoperitoneum during Robotic Partial Nephrectomy.
  Interventions: Device: SurgiQuest AirSeal Insufflation System (AIS)
- AIS @ 15mmHg pressure (Active Comparator): SurgiQuest AirSeal insufflation System (AIS) set at 15 mmHg pressure for the management of pneumoperitoneum during Robotic Partial Nephrectomy.
  Interventions: Device: SurgiQuest AirSeal Insufflation System (AIS)
- CIS @ 15mmHg pressure (Active Comparator): Conventional Insufflation System (CIS) set at 15mmHg pressure for the management of pneumoperitoneum during Robotic Partial Nephectomy.
  Interventions: Device: Conventional Insufflation System (CIS)

INTERVENTIONS:
Device: SurgiQuest AirSeal Insufflation System (AIS) — Comparison between Conventional Insufflation System (CIS) and the SurgiQuest AirSeal Insufflation System (AIS) at similar pressures (15mmHg) and the SurgiQuest AirSeal at 12mmHg.
  Arms: AIS @ 12mmHg pressure; AIS @ 15mmHg pressure
Device: Conventional Insufflation System (CIS) — Comparison between Conventional Insufflation System (CIS) and the SurgiQuest AirSeal Insufflation System (AIS) at similar pressures (15mmHg) and the SurgiQuest AirSeal at 12mmHg.
  Arms: CIS @ 15mmHg pressure

SUMMARY:
A MULTI-CENTER, PROSPECTIVE, RANDOMIZED, CONTROLLED STUDY TO EVALUATE PHYSICIAN PREFERENCE RELATED TO THE USE OF THE SURGIQUEST AIRSEAL INSUFFLATION SYSTEM (AIS) VS. CONVENTIONAL INSUFFLATION SYSTEMS (CIS) FOR THE MANAGEMENT OF PNEUMOPERITONEUM DURING ROBOTIC PARTIAL NEPHRECTOMY

DETAILED DESCRIPTION:
A prospective, randomized, controlled multi-center clinical Study designed to evaluate Physician Preference related to the use of the SurgiQuest AirSealTM Insufflation System (AIS) vs. Conventional Insufflation Systems (CIS) for the Management of pneumoperitoneum during Robotic Partial Nephrectomy. Subjects will be randomized in a 1:1:1 treatment device to control ratio into one of three (3) different study arms: 1) AIS @ 12mmHg pressure, 2) AIS @ 15mmHg pressure, and 3) CIS @ 15mmHg pressure. 189 randomized subjects distributed in three arms of 63 patients. The three study sites are targeted to enroll 63 patients each, 21 patients in each of the three (3) study arms. It is expected that this will take up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for an elective, non-emergent robotic partial nephrectomy;

Exclusion Criteria:

Subjects will be excluded from participating in this Study if they meet any of the following criteria prior to initiation of the endoscopic procedure 1.Advanced refusal of blood transfusion, if necessary; 2.Active systemic or cutaneous infection or inflammation; 3 Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids; 4.Uncontrolled diabetes mellitus 5.Known, significant history of bleeding diathesis, coagulopathy, von Willebrand's disease or current platelet count < 100,000 cells/mm3, baseline INR ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours); 6.Severe co-existing morbidities having a life expectancy of less than 30 days; 7.Currently involved in any other investigational clinical Studies; 8.Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%; 9.Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating; 10.Extreme morbid obesity (BMI greater than 45 kg/m2) or underweight (BMI less than 20 kg/m2); 11. Patients presenting with Ascites

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Rate of insufflation device related subcutaneous emphysema (SCE) at 2 hours | 2 hours post procedure
  Rate of insufflation device related subcutaneous emphysema(SCE)
Rate of insufflation device related subcutaneous emphysema (SCE) at 4 hours | 4 hours post procedure
  Rate of insufflation device related subcutaneous emphysema(SCE)
Rate of insufflation device related subcutaneous emphysema (SCE) at 8 hours | 8 hours post procedure
  Rate of insufflation device related subcutaneous emphysema(SCE)
Rate of insufflation device related subcutaneous emphysema (SCE) at 12 hours | 12 hours post procedure
  Rate of insufflation device related subcutaneous emphysema(SCE)
Rate of insufflation device related subcutaneous emphysema (SCE) at 24 hours | 24 hours post procedure
  Rate of insufflation device related subcutaneous emphysema(SCE)

SECONDARY OUTCOMES:
Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) required pain medication, measured with Visual Analogue Scale (VAS) | 2, hours post procedure
  Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) measured with Visual Analogue Scale (VAS), required pain medication
Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) required pain medication, measured with Visual Analogue Scale (VAS) | 4 hours post procedure
  Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) measured with Visual Analogue Scale (VAS), required pain medication
Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) required pain medication, measured with Visual Analogue Scale (VAS) | 8 hours post procedure
  Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) measured with Visual Analogue Scale (VAS), required pain medication
Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) required pain medication, measured with Visual Analogue Scale (VAS) | 12 hours post procedure
  Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) measured with Visual Analogue Scale (VAS), required pain medication
Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) required pain medication, measured with Visual Analogue Scale (VAS) | 24 hours post procedure
  Rate of Pneumothorax, Pneumomediastinum, Post op pain (general/shoulder) measured with Visual Analogue Scale (VAS), required pain medication

CONTACTS AND LOCATIONS:
Overall Officials: James Porter, MD, Principal Investigator — Swedish Medical Center, Seattle , WA
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Swedish Medical Center, Seattle, Washington